CLINICAL TRIAL: NCT02139007
Title: Effectiveness of DiscontinuinG bisphosphonatEs Study: R21 Pilot Study
Acronym: EDGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F120404006
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuation Arm (Active Comparator): Alendronate continuation arm
  Interventions: Drug: Alendronate
- Discontinuation Arm (Active Comparator): Alendronate discontinuation arm
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
This is a pilot study evaluating the recruitment strategies for sites and patients, data collection instruments, follow-up procedures, administrative processes, and the proposed management strategy for the future large scale national trial.

ELIGIBILITY:
Inclusion Criteria:

1.Females 65+

2.3+ years of alendronate (Fosamax/Binosto) use

3. Valid social security number

Exclusion Criteria:

1. History of any other metabolic bone condition, such as Paget Disease of Bone
2. Currently receiving treatment for ongoing cancer, excluding non-melanoma skin cancer.
3. Has significant underlying illness that would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 3 years)?
4. HIV positive
5. Involved in a conflicting (investigational drug) clinical trial

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Saag, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sites were selected from 2 practice based research networks based upon self-reporting having a large number of women ≥ 65 years of age with a current alendronate prescription. Enrolled patient participants were randomized to continue or discontinue their current prescription. No drug was provided.
Pre-assignment Details: Period 1 refers to the study site recruitment period for the 9 sites that participated in the study. Period 2 refers to the patient recruitment period for the study. Randomization to treatment assignment was at the patient level. Sites recruited patient participants to both arms of the study. Two sites failed to enroll participants in either arm.
Groups:
- Continuation Arm: Alendronate continuation arm
  Participants were randomized to continue their current alendronate prescription at prescribed dose.
- Discontinuation Arm: Alendronate discontinuation arm
  Participants were randomized to stop taking their current alendronate prescription.
Period: Study Site Recruitment
Arm/Group | Continuation Arm | Discontinuation Arm
Started | 4 | 5
Completed | 1 | 1
Not Completed | 3 | 4
Period: Patient Participant Recruitment
Arm/Group | Continuation Arm | Discontinuation Arm
Started | 13 | 14
Completed | 11 | 13
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuation Arm | Discontinuation Arm | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.4 (6.7) | 74.5 (5.9) | 74.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Previous History of Fracture [Count of Participants; unit: Participants] | 5 | 5 | 10
Duration of Alendronate Use [Mean (Standard Deviation); unit: Years] | 4.8 (2.1) | 5.3 (3.1) | 5.1 (17)

OUTCOME MEASURES:

1. Primary Outcome: All Study Sites--Length of Contracting Procedures
Description: Mean time Between Clinical Site Recruitment and Contract Execution
Time Frame: Length of time Between Clinical Site Recruitment and Contract Execution
Population: Nine sites from six states (AL, CO, NM, CT, CA, and PA) participated in this pilot study.
Measure: Mean (Standard Deviation); unit: Months
Units Other Than Participants: Sites
Groups:
- All Study Sites -- Contracting Procedures: The duration of time from execution of contracts, IRB approval, and to participant recruitment is potential contributor to overall suboptimal recruitment in clinical research. In this pilot study we measured the mean duration of administrative procedures for sites to the first patient enrolled. .
Arm/Group | All Study Sites -- Contracting Procedures
Number analyzed (Participants) | 9
Number analyzed (Sites) | 9
Months | 3.4 (2.3)

2. Primary Outcome: All Study Sites--Length of Time to Site IRB Approval
Description: Mean time to gain site IRB approval
Time Frame: Length of time to site IRB approval
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Sites
Groups:
- All Study Sites --IRB Approval: The duration of time from execution of contracts, IRB approval, and to participant recruitment is potential contributor to overall suboptimal recruitment in clinical research. In this pilot study we measured the mean duration of administrative procedures for sites to the first patient enrolled. .
Arm/Group | All Study Sites --IRB Approval
Number analyzed (Participants) | 9
Number analyzed (Sites) | 9
Days | 13.9 (4.1)

3. Primary Outcome: All Study Sites-Length of Time to 1st Participant Enrolled
Description: Mean time from study initiation to 1st participant enrolled.
Time Frame: Length of time t for sites to recruit/enroll 1st participant
Population: For sites enrolling at least one patient, the average (SD) time from contract execution to the first patient recruited.
Measure: Mean (Standard Deviation); unit: Months
Units Other Than Participants: Sites
Groups:
- All Study Sites-Initiation to the First Participant Recruited: study initiation to the first participant recruited
Arm/Group | All Study Sites-Initiation to the First Participant Recruited
Number analyzed (Participants) | 9
Number analyzed (Sites) | 9
Months | 5.0 (3.0)

4. Secondary Outcome: Clinical Fracture Rate
Description: Patient reported fracture rate at 6 months following enrollment via survey.
Time Frame: Baseline to 6 months following enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Continuation Arm: Alendronate continuation arm
  Alendronate
- Discontinuation Arm: Alendronate discontinuation arm
  Alendronate
Arm/Group | Continuation Arm | Discontinuation Arm
Number analyzed (Participants) | 11 | 13
Participants | 0 | 0

5. Secondary Outcome: Atypical Femoral Fracture
Description: Patient reported fracture rate at 6 months after enrollment via follow-up survey
Time Frame: Baseline to 6 months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Arm | Discontinuation Arm
Number analyzed (Participants) | 11 | 13
Participants | 0 | 0

6. Secondary Outcome: Osteonecrosis of the Jaw
Description: Patients self report diagnoses of osteonecrosis of the jaw 6 months post enrollment via follow-up survey .
Time Frame: Baseline to 6 months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Arm | Discontinuation Arm
Number analyzed (Participants) | 11 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 6 months following enrollment
Arm/Group | Continuation Arm | Discontinuation Arm
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes